CLINICAL TRIAL: NCT01598441
Title: Multi-centre, Randomized Study of Iloprost Inhaled in Preventing and Treating Reactive Pulmonary Hypertension (RPH) and Pulmonary Hypertensive Crisis (PHC) After Repair of Congenital Heart Diseases (CHD)
Brief Title: Multicenter Study of Iloprost Inhaled in Pulmonary Hypertension After Repair of Congenital Heart Diseases (CHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Cardiothoracic Surgical Group of Chinese Society of Pediatric Surgery (Unknown)
Responsible Party: Principal Investigator, Xu Zhuoming, Director of ICU, Department of thoracic and cardiovascular surgery, Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCMCIRB-201127
Record Dates: First submitted 2012-05-06; First posted 2012-05-15 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension, pulmonary hypertensive crisis
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iloprost (Experimental): Iloprost nebuliser solution 500 ng/kg inhaled
  Interventions: Drug: iloprost nebuliser solution
- distilled water (Placebo Comparator): aerosolized distilled water 1-2 ml
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: iloprost nebuliser solution — Iloprost nebuliser solution 500 ng/kg inhaled(10 min recommended) q3h for 2 days
  Other Names: Ventavis
  Arms: iloprost
Drug: distilled water — 1-2 ml aerosolized distilled water inhalation per session
  Other Names: Treeful
  Arms: distilled water

SUMMARY:
This study was designed to investigate treatment of postoperative pulmonary hypertension by iloprost inhalation in children with congenital heart defects. It was a controlled single-blind randomized multi-center prospective study in order to explore the efficacy of this method in the treatment and prevention of pediatric pulmonary hypertension after corrective open-heart surgery for congenital heart defects.

DETAILED DESCRIPTION:
Primary objectives:

1. To evaluate the effect of iloprost inhaled on postoperative PH after biventricular repair for CHD.
2. To verify the benefits of iloprost inhaled in improving the hemodynamics after biventricular repair for CHD.

Secondary objectives:

1. To investigate the preventive effect of iloprost inhaled on the life-threatening PHC occurring immediately after complex congenital heart surgery or occurring just after weaning off cardiopulmonary bypass.
2. To explore the potential of iloprost inhaled to reduce the early mortality after PHC and to decrease the use of ECMO/VAD.

ELIGIBILITY:
Inclusion Criteria:

* CHD children who have associated PH risk factors and have accepted biventricular repair
* Pp/Ps >= 0.75 (before surgery) or Pp/Ps >= 0.5 (after surgery)

Exclusion Criteria:

* severe mitral stenosis
* obstructive drainage of pulmonary veins
* platelet count < 50,000,000,000/L & obvious bleeding

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The total incidence of RPH, PHC or death | within 48 hours after surgery
  The primary effective endpoints are reached when any individual components of the primary composite endpoint occur:
  * RPH lasting for more than 30 mintues; or
  * PHC at any time; or
  * death

SECONDARY OUTCOMES:
Change from base line of pulmonary hemodynamic measurements | within 48 hours after surgery
  * Pp/Ps
  * NYHA class function
  * SvO2
  * PAO2

CONTACTS AND LOCATIONS:
Overall Officials: Zhuomin Xu, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Guangzhou Children's Hospital, Guangzhou, Guangdong
  - Wuhan Asia Hear Hospital, Wuhan, Hubei
  - Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center, Shanghai